CLINICAL TRIAL: NCT03653312
Title: Neuromuscular Electrical Stimulation in Acute Ischemic Stroke
Acronym: NESA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-80-2015
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Stroke; Neuromuscular Electrical Stimulation; Exercise
Keywords: Ischemic Stroke; Neuromuscular electrical stimulation; Activities of daily living; Patient reported outcome; Fugl Meyer
MeSH Terms: conditions — Ischemic Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel group, assessor blinded, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: One blinded outcome assessor (physiotherapists) will perform measurements of functional capacity, patient reported outcome, and cognition. Statistical analysis will be performed by a blinded statistician and a blinded interpretation of the results will be performed before breaking the randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES (Active Comparator): 2 weeks (weekdays) of Neuromuscular Electrical Stimulation of the paretic lower limb during exercise.
  Each exercise session will last for 12 minutes and will consist of either walk or sit and raise from a chair.
  Interventions: Device: NMES
- training (No Intervention): Participants will undergo 2 weeks of exercise every weekday. Each exercise session will last for 12 minutes and will consist of either walk or sit and raise from a chair.

INTERVENTIONS:
Device: NMES — Neuromuscular electrical stimulation of the paretic lower limb during exercise
  Arms: NMES

SUMMARY:
The purpose of the study is to examine the added effect of NeuroMuscular Electric Stimulation (NMES) in addition to exercise therapy in the acute phase of ischemic stroke.

This randomized controlled trial includes 50 patients allocated to either control or intervention.

The inclusion, test, training and re-test will be provided during the first 14 days after ictus, starting day 1 or 2 after ictus and a follow-up at day 90.

The exercise training with external NMES is done with the patient every weekday for 12 minutes.

DETAILED DESCRIPTION:
Stroke is the third most cause of disability in adults over 65 years of age worldwide. In 2008, 30.7 million people had survived a stroke. Every year, there are about 14,000 new cases of stroke in Denmark and the number is expected to rise with about 40% by 2035, due to the increasing population of elderly. Stroke survivors have the worst odds of reporting severe disability and the greatest variety of individual domains of disability compared to a range of other diseases. Therefore, these patients have essential rehabilitation needs. Little is known about who will benefit from functional interventional rehabilitation and what kind of intervention is best.

The purpose of the study is to examine the added effect of NeuroMuscular Electric Stimulation (NMES) in addition to exercise therapy in the acute phase of ischemic stroke.

This RCT includes 50 patients allocated to either control or intervention. The inclusion, test, training and re-test will be provided during the first 14 days after ictus, starting day 1 after ictus and a follow-up at day 90.

The exercise training with external NMES is done with the patient every weekday for 12 minutes.

If NMES increases functionality in acute stroke patients it would mean a greater degree of independence for individual patients and thus have the potential to improve on a major problem for society.

By combining comorbidity, stroke severity, and other demographic data it might be possible to get a greater knowledge about who will benefit from the intervention and early rehabilitation and that will be the a step towards "personalized medicine" in stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic apoplexy and paresis in lower extremity, verified with picture diagnosis (CT/MR) or clinically diagnosed.
* Leg palsy equalizes 2-4
* Modified Ranking Scale(mRS) =0-1
* Cognitive function adequate to participate

Exclusion Criteria:

* Patients with dementia and/or malign diseases
* Pregnancy
* Epilepsy
* Total loss of sensation
* Pacemaker
* Previous or current blood clot in the leg
* Untreated depression
* Untreated alcohol or drug abuse
* Untreated hypertension
* Heart disease which limits function

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The six Minute-Walk Test | Primary endpoint: Change from baseline to 3 months. Secondary endpoint: Change from baseline to 2 weeks.
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.

SECONDARY OUTCOMES:
Fugl Meyer Assessment | Primary endpoint: Change from baseline to 3 months. Secondary endpoint: Change from baseline to 2 weeks.
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia
Sit to stand | Primary endpoint: Change from baseline to 3 months. Secondary endpoint: Change from baseline to 2 weeks.
  Sit-to-stand is a mechanically demanding task demanding task
Timed Up and Go | Primary endpoint: Change from baseline to 3 months. Secondary endpoint: Change from baseline to 2 weeks.
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
EuroQOL 5 domain | Change from day 14 post ictus to day 90 post ictus.
  A self-reported outcome measure of health-related quality of life, covering 5 dimensions (movement, personal care, everyday activities, pain/discomfort and anxiety/depression). Is translated and validated for use in a Danish population.
10 meter walk test | Primary endpoint: Change from baseline to 3 months. Secondary endpoint: Change from baseline to 2 weeks.
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a 10 meter distance.
Montreal Cognitive Assessment (MoCA) | Change from day 14 post ictus to day 90 post ictus.
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Becks Depression Inventory | Change from day 14 post ictus to day 90 post ictus.
  Becks Depression Inventory is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression
Guralnik | Primary endpoint: Change from baseline to 3 months. Secondary endpoint: Change from baseline to 2 weeks.
  Balance test assessed by the ability to stand for 10 seconds without support in each of the following positions: total feet, semitandem and full tandem

CONTACTS AND LOCATIONS:
Overall Officials: Troels Wienecke, MD, PhD, Study Director — Department of Neurology, Zealand University Hospital, University of Copenhagen, Roskilde, Denmark; Henriette Busk, PT, Principal Investigator — Dept. of Neurology, Zealand University Hospital, and Department of Physiotherapy and Occupational Therapy, Naestved-Slagelse-Ringsted Hospital, Copenhagen University; Søren T Skou, PT, PhD, Study Chair — University of Southern Denmark and Naestved-Slagelse-Ringsted Hospitals; Gert Kwakkel, Study Chair — Dept. Rehabilitation Medicine, VU University Medical Center, Amsterdam, The Netherlands
Locations (1):
- Department of Neurology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03653312/SAP_000.pdf